CLINICAL TRIAL: NCT00030888
Title: A Phase 2 Study Of UCN-01 In Advanced Renal Cell Carcinoma
Brief Title: UCN-01 in Treating Patients With Advanced or Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069208; UCSF-NCI-5522; NCI-5522
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — 7-hydroxystaurosporine

INTERVENTIONS:
Drug: 7-hydroxystaurosporine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of UCN-01 in treating patients who have unresectable stage III or stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of UCN-01, in terms of time to objective progression, in patients with stage IV or unresectable stage III renal cell carcinoma.
* Determine the objective response rate in patients treated with this drug.

OUTLINE: Patients receive UCN-01 IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 21-61 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV or unresectable stage III renal cell carcinoma

  * Metastatic disease must be amenable to biopsy or appropriate for nephrectomy before study therapy
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known prior or concurrent CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of clinically significant coronary artery disease
* No symptomatic cardiac dysfunction
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary:

* No symptomatic pulmonary dysfunction

Other:

* No prior allergic reactions to compounds of similar chemical or biological composition to UCN-01
* No other uncontrolled concurrent illness
* No active or ongoing infection
* No known immune deficiency
* No psychiatric illness or social situation that would preclude study compliance
* No insulin-dependent diabetes mellitus
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No prior mediastinal radiation

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior nephrectomy

Other:

* No more than 2 prior systemic therapies for metastatic renal cell carcinoma
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Rini, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California